CLINICAL TRIAL: NCT02872376
Title: Clinical Burden of Anemia in Inflammatory Bowel Disease: Role of Iron Deficiency And Iron Replacement Therapy, Observational Study (RIDART-1)
Brief Title: Clinical Burden of Anemia in Inflammatory Bowel Disease (RIDART1)
Acronym: RIDART-1
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Antonio Di Sabatino, Associate Professor of Internal Medicine, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: RIDART-I
Record Dates: First submitted 2016-08-09; First posted 2016-08-19 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Anemia
Keywords: Anemia; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Anemia; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Anemic: Anemic patients

SUMMARY:
Anemia is the most common extraintestinal manifestation of IBD, occurring in 6 to 74 percent of patients. Most cases of anemia in IBD are due to iron deficiency (IDA) and to anemia of inflammation (AI). Although the ECCO diagnostic criteria for IDA are simple, and iron supplementation represents a cheap and usually effective treatment, many IBD patients with IDA are not properly treated. The inconsistent adherence, by many physicians, to treatment guidelines for IDA in IBD is often motivated by the belief that mild to moderate degrees of anemia may not have a significant impact on the patient's quality of life or do not represent the main clinical problem of the patient, that oral iron supplementation may adversely affect disease activity, and that parenteral iron administration may cause severe side effects. On this basis, we aim to perform a longitudinal, prospective, observational study whose main objective is the determination of the prevalence of anemia in IBD patients in Italy. Secondary objectives of the study are a) to investigate the pathogenesis of anemia in IBD, with a particular focus on the differential diagnosis between IDA and AI, and how disease activity, extension or behavior influence the relative frequency of IDA and AI; b) to verify the adherence to ECCO guidelines for the treatment of IDA in IBD (the proportion of patients with IDA that receive adequate iron supplementation); c) to administer dedicated questionnaires to the patients in order to measure the influence of anemia on fatigue and quality of life among IBD patients.

DETAILED DESCRIPTION:
BACKGROUND

Anemia is the most common extraintestinal manifestation of IBD, occurring in 6 to 74 percent of patients. This wide range in the prevalence of anemia is related to differences in study design, in the criteria used to define anemia and to the increasing awareness of anemia in these patients. According to a recent meta-analysis of European studies involving 2192 IBD patients, the overall prevalence of anemia in Europe was 27%, ulcerative colitis patients being less likely to develop anemia than those with Crohn's disease. Therefore, anemia represents a significant clinical and social burden in IBD management; this is more evident in southern Europe where the prevalence of anemia is close to 40%. Most cases of anemia in IBD are due to iron deficiency (IDA) and to anemia of inflammation (AI). Guidelines concerning the diagnosis and treatment of IDA in IBD have been published by the European Crohn's and Colitis Organisation. According to present guidelines iron supplementation should be started when IDA is present or even in the presence of iron deficiency without anemia. A meta-analysis of iron supplementation studies in IBD-associated IDA found that intravenous iron is more effective and better tolerated than oral iron supplementation, but the sample size of the included studies was small; absolute indications for intravenous iron include severe anemia (haemoglobin <10.0 g/dL) and intolerance or inadequate response to oral iron.

Although the ECCO diagnostic criteria for IDA are simple, and iron supplementation represents a cheap and usually effective treatment, many IBD patients with IDA are not properly treated. The inconsistent adherence, by many physicians, to treatment guidelines for IDA in IBD is often motivated by the belief that mild to moderate degrees of anemia may not have a significant impact on the patient's quality of life or do not represent the main clinical problem of the patient, that oral iron supplementation may adversely affect disease activity, and that parenteral iron administration may cause severe side effects.

RATIONALE

In order to improve the diagnostic and therapeutic work-up of anemia in IBD, it is necessary to precisely define the prevalence and pathogenesis of anemia in the Italian IBD population and gain informations about how anemic patients, particularly those with IDA, are usually managed and followed-up. In addition, since IDA and AI are the most common forms of anemia in IBD, and both mechanisms often concur to the pathogenesis of anemia in the same subject, stringent diagnostic criteria to distinguish the three conditions (IDA, AI and coexistence of IDA and AI) are urgently needed. The differential diagnosis between IDA and AI is often difficult since inflammation modifies serum ferritin and transferrin saturation (TfSat) that become unreliable as indicators of iron status. Recently, serum hepcidin concentration has been identified as a new index of iron status that can be useful to differentiate IDA and AI in IBD. Hepcidin, a peptide produced by the liver in response to increased iron stores, inflammation and reduced erythropoietic activity, is the master regulator of body iron homeostasis and acts by inhibiting iron absorption and iron release from hepatocytes and macrophages to plasma. The potential role of serum hepcidin determination as a diagnostic tool in the differential diagnosis of anemia in IBD and in other inflammatory diseases must be clearly defined. The investigation of these topics is important since a more accurate pathogenetic diagnosis of anemia in IBD, while preventing the useless and potentially harmful treatment of AI with iron supplementation, might allow the identification and appropriate treatment of IDA patients in the presence of inflammation.

STUDY DESIGN

We will perform a longitudinal, prospective, observational study whose aim is the determination of the prevalence and pathogenesis of anemia in IBD patients. Anemia is defined according to WHO criteria: Hb <13.0 g/dL for males and Hb <12 g/dL for females. Anemia work-up should be initiated whenever Hb concentration is below normal and will include the determination of the laboratory parameters reported in the CRF. A serum ferritin <100 µg/L and transferrin saturation <20% are required for the diagnosis of isolated IDA and for the association of IDA and inflammation. We plan to involve at least 60 IG-IBD Centers in this observational study. We expect to include 2000 anemic patients in the study; approximately 80 to 90% of these patients will have some form of iron deficiency and/or AI. This will allow to evaluate differences in prevalence of IDA and AI according to gender, age, diagnosis, time from diagnosis, presence of inflammation, activity, extension and behaviour of the disease, and to evaluate variables associated with type and severity of anemia in both univariate and multivariate analysis. Expected duration of subject participation to both the observational and the therapeutic trials will be 24 weeks; all anemic patients recruited in the study will undergo screening to investigate the mechanism of anemia, and follow-up evaluation will be performed at weeks 4, 12 and 24. At follow-up, informations about the treatment of anemia, fatigue and quality of life must be collected.

OBJECTIVES

Primary endpoint of this observational study is to determine the prevalence of anemia in Italian patients with IBD. Secondary objectives of the study are a) to investigate the pathogenesis of anemia in IBD, with a particular focus on the differential diagnosis between IDA and AI, and how disease activity, extension or behavior influence the relative frequency of IDA and AI; b) to verify the adherence to ECCO guidelines for the treatment of IDA in IBD (the proportion of patients with IDA that receive adequate iron supplementation); c) to administer dedicated questionnaires to the patients in order to measure the influence of anemia on fatigue and quality of life among IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged 18 years and over
* Have IBD and anemia

Exclusion Criteria:

- IBD patients without anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease and anemia
Sampling Method: Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ratio of the number of anemic patients over the number of patients screened for anemia | 12 months
  The primary outcome will be computed as the ratio of the number of anemic patients over the number of patients screened for anemia together with its 95% confidence interval

SECONDARY OUTCOMES:
Ratio between the number of patients with IDA or with AI over the total number of anemic patients | 12 months
  Relative prevalence of IDA and AI in IBD will be computed as the ratio between the number of patients with IDA or with AI over the total number of anemic patients
IBDQ | 12 months
  Influence of anemia on quality of life among IBD patients
Number of hospitalizations in anemic patients | 12 months
  Influence of anemia on hospitalization rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Derived] Bergamaschi G, Castiglione F, D'Inca R, Astegiano M, Fries W, Milla M, Ciacci C, Rizzello F, Saibeni S, Ciccocioppo R, Orlando A, Bossa F, Principi M, Vernia P, Ricci C, Scribano ML, Bodini G, Mazzucco D, Bassotti G, Riegler G, Buda A, Neri M, Caprioli F, Monica F, Manca A, Villa E, Fiorino G, Comberlato M, Aronico N, Della Corte C, Caccaro R, Gionchetti P, Giuffrida P, Iovino P, Lenti MV, Mengoli C, Pellegrini L, Pieraccini A, Ribaldone D, Testa A, Ubezio C, Viola A, Vecchi M, Klersy C, Di Sabatino A. Prevalence, Pathogenesis and Management of Anemia in Inflammatory Bowel Disease: An IG-IBD Multicenter, Prospective, and Observational Study. Inflamm Bowel Dis. 2023 Jan 5;29(1):76-84. doi: 10.1093/ibd/izac054. PMID 35366312
- Available data/document: Study Protocol — https://sites.google.com/site/ridartstudy/
- Available data/document: Informed Consent Form — https://sites.google.com/site/ridartstudy/